CLINICAL TRIAL: NCT03698565
Title: Evaluation of the Analgesia Nociception Index and Videopupillometry to Predict a Child's Post-tonsillectomy Morphine Prescription
Acronym: ENIGME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RC17_0109 (ENIGME)
Record Dates: First submitted 2018-09-24; First posted 2018-10-09 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative
Keywords: Pain Postoperative; Tonsillectomy; Analgesia Nociception Index; Pupillary Index Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PPI and ANI measurements (Experimental): The intervention is the nerve stimulation of the ulnar nerve for evaluation / realization of PPI by videopupillometry.
  The realization of PPI and ANI measurements is carried out at the end of the surgical procedure, it implies a maintenance of the anesthesia for approximately 5 additional minutes.
  Interventions: Other: Nerve stimulation of the ulnar nerve

INTERVENTIONS:
Other: Nerve stimulation of the ulnar nerve — The intervention is the nerve stimulation of the ulnar nerve for evaluation / realization of PPI by videopupillometry.
  The realization of PPI and ANI measurements is carried out at the end of the surgical procedure, it implies a maintenance of the anesthesia for approximately 5 additional minutes.

SUMMARY:
Some surgeries, such as tonsillectomies, are particularly painful postoperatively because they are not very accessible to a complementary technique of loco-regional anesthesia and require the use of opioids in the postoperative period.

The use of opioids, in combination with usual analgesics, is common after this surgery. However, some risks are associated with the use of morphine in children, including more frequent respiratory distress, nausea and vomiting, and can cause hemorrhagic complications and lengthen the duration of hospitalization. Decreasing the consumption of morphine drugs is therefore a real challenge.

Although there is no randomized controlled study on the use of standard analgesics with or without morphine to date, a number of studies suggest that the use of morphine should not be systematic after a surgery.

The need for opioids after tonsillectomy as well as the level of pain vary between patients. Some teams use morphine at the end of general anesthesia to prevent pain on waking and others use it only if needed, once the child is awake.

Pain assessment scales are used in the Post-interventional Monitoring Room (PIMR) to adapt these analgesic therapies according to the intensity of pain. One of the validated and frequently used scales in pediatric PIMR is FLACC (Face Legs Activity Cry Consolability). Monitoring tools are also available to evaluate the quality of intraoperative analgesia in unconscious children :

* the analysis of the pupillary variation in response to a painful stimulus by videopupillometry,
* and the ANI (Analgesia Nociception Index) which consists of estimating the sympathetic-parasympathetic balance by a complex analysis of cardiac rhythm variability.

These two types of monitoring could predict which children will require post-operative morphine treatment.

To date, no study has demonstrated the relationship between videopupillometry and postoperative morphine consumption. The average ANI has already been evaluated in children as correlated with FLACC but both monitoring devices have never been compared for a predictive purpose.

The investigators hypothesize that the use of the PPI® (Pain Pupillary Index) scale of Algiscan® and the average ANI measured by the PhysioDoloris® monitor in children still sedated at the end of the intervention could have a prognostic value on post-operative morphine prescription.

ELIGIBILITY:
Inclusion Criteria:

* Any child for whom tonsillectomy is programmed ≥ 2 years and up to 7 years inclusive
* Consent written and signed by at least one holder of exercise of parental authority

Exclusion Criteria:

* Eye disease
* Cardiac pathology
* Neurological pathology
* Chronic opioid treatment
* Any treatment interfering with the autonomic nervous system
* Any contraindication to NSAIDs

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Prognostic value of the Pupillary Index Pain ® measured at the end of the surgical intervention | Day 0 (End of the surgery)
  Presence or absence of a morphine prescription during the SSPI.
Prognostic value of the average Analgesia Nociception Index measured at the end of the surgical intervention | Day 0 (End of the surgery)
  Presence or absence of a morphine prescription during the SSPI.

SECONDARY OUTCOMES:
Correlation between Analgesia Nociception Index measured and maximum score obtained at FLACC scale | Day 1 (Leaving the Post-interventional Monitoring Room)
  The correlation coefficient of Pearson or Spearman between the Analgesia Nociception Index measured by the PhysioDoloris® monitor at the end of the surgical intervention and the maximum score obtained at the FLACC scale during the stay in the Post-interventional Monitoring Room.
Correlation between Pain Pupillary Index measured and maximum score obtained at FLACC scale | Day 1 (Leaving the Post-interventional Monitoring Room)
  The correlation coefficient of Pearson or Spearman between the Pupillary Index ® Pain measured by Algiscan at the end of the surgical intervention and the maximum score obtained at the FLACC scale during the stay in the Post-interventional Monitoring Room.
Correlation between variation of the pupillary diameter measured and maximum score obtained at FLACC scale | Day 1 (Leaving the Post-interventional Monitoring Room)
  The correlation coefficient of Pearson or Spearman between the change in pupillary diameter measured by Algiscan® at the end of the surgical intervention and the maximum score obtained at the FLACC scale during the stay in the Post-interventional Monitoring Room.

CONTACTS AND LOCATIONS:
Overall Officials: Charles HODLER, PH, Principal Investigator — University Hospital, Limoges
Locations (1):
- University Hospital, Limoges, France

REFERENCES:
- [Background] Evrard B, Lefebvre C, Spiry P, Hodler C, Chapellas C, Youssef B, Gauthier F, Marais L, Labrunie A, Douchez M, Senges P, Cros J, Nathan-Denizot N. Evaluation of the Analgesia Nociception Index and videopupillometry to predict post-tonsillectomy morphine requirements in children: a single-centre, prospective interventional study. BJA Open. 2022 Jul 31;3:100024. doi: 10.1016/j.bjao.2022.100024. eCollection 2022 Sep. PMID 37588574